CLINICAL TRIAL: NCT01921686
Title: Dilation of Intercellular Spaces as Morphological Markers of Gastroesophageal Reflux Disease (GERD)In Children
Brief Title: Morphological Markers of Gastroesophageal Reflux Disease (GERD)
Status: Active, not recruiting | Type: Observational
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Eric Chiou, Assistant Professor, Baylor College of Medicine
Other Study IDs: H-28604
Record Dates: First submitted 2013-08-09; First posted 2013-08-13 (Estimated); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Eosinophilic Esophagitis; Gastroesophageal Reflux Disease
Keywords: Eosinophil; Reflux; Esophagus; Food allergy; Trouble Swallowing; Pediatrics; Healthy Volunteers
MeSH Terms: conditions — Eosinophilic Esophagitis; Gastroesophageal Reflux; Food Hypersensitivity; Deglutition Disorders | interventions — Specimen Handling; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Three esophageal biopsy samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Gastroesophageal Reflux Disease (GERD): History of troublesome symptoms (e.g. heartburn, chest pain, acid regurgitation) secondary to reflux of gastric contents at least three times per week
  AND, At least one of the following:
  * Mucosal breaks on endoscopy (at least Grade-A esophagitis based on Los Angeles classification)
  * Abnormal pH index (pH less than 4 for greater than 6% of study)
  * Abnormal MII-pH (greater than 73 episodes of total reflux per 24 hours)
  Interventions: Other: Sample collection and Questionnaire
- Eosinophilic Esophagitis (EoE): * History of troublesome esophageal symptoms (e.g. dysphagia, food impaction, vomiting, upper abdominal or chest pain)
  * Greater than or equal to 15 eosinophils in at least one high powered field (HPF) from distal OR proximal esophageal biopsy
  * Lack of histological response to 6-8 weeks of high dose Proton Pump Inhibitor (PPI) OR negative pH probe (pH less than 4 for less than 6% of study). Subjects with greater than 15 eosinophils/HPF and abnormal pH results may have an overlap syndrome and will be excluded from the primary analysis.
  Interventions: Other: Sample collection and Questionnaire
- Control: Patients with no history of troublesome esophageal symptoms or esophageal disease AND normal esophagoscopy (for example, patients undergoing evaluation for chronic abdominal pain, inflammatory bowel disease, celiac disease).
  Interventions: Other: Sample collection and Questionnaire

INTERVENTIONS:
Other: Sample collection and Questionnaire — This is an observational biospecimen collection and questionnaire study. The subjects will be asked to complete a symptom questionnaire at screening visit. In addition, 3 esophageal biopsy samples will be taken to conduct laboratory analyses.

SUMMARY:
The purpose of this project is to learn more about a new and promising way to diagnose acid reflux disease using a very high-powered microscope. This special microscope provides much finer detail than typical microscopes previously used for diagnosing reflux, and may help doctors to better identify children with acid reflux.

DETAILED DESCRIPTION:
This will be a prospective case control study. Children between the ages of 8 and 18 with suspected gastroesophageal reflux disease (GERD) or eosinophilic esophagitis (EoE) based on symptom criteria and who have been scheduled for esophagogastroduodenoscopy (EGD) by their primary gastroenterologist will be recruited.

Children who do not have any history of esophageal disease or esophageal symptoms and are scheduled for EGD for other clinical indications (e.g. rule out celiac disease) by their primary gastroenterologist will be recruited and act as controls. Control subjects will also be given the opportunity to undergo esophageal MII-pH monitoring as part of their medical evaluation, but will not be excluded from analysis should they opt out of this part of the study.

For all subjects, in addition to endoscopic evaluation, biopsies of the distal esophagus will be obtained for routine light microscopy (standard histology sample) as well as Transmission Electron Microscopy (TEM) analysis to determine the presence and magnitude of dilated intercellular spaces (DIS), and immunoblotting for e-cadherin cleavage

ELIGIBILITY:
Inclusion Criteria for GERD or EoE Subjects:

* Children between the ages of 8-18 years
* Suspected diagnosis of GERD or EoE based on symptom criteria
* Able to tolerate upper endoscopy examination with biopsies

Inclusion Criteria for Control Subjects:

* Children between the ages of 8-18
* Scheduled for EGD for clinical indications
* No history of esophageal disease of esophageal symptoms
* Able to tolerate upper endoscopy examination with biopsies

Exclusion Criteria for GERD or EoE Subjects:

* History of Barrett's esophagus
* Previous esophageal or gastric surgery
* History of congenital defect/malformation of the esophagus
* Diagnosis of Crohn disease

Exclusion Criteria for Control Subjects:

* Symptoms of GERD or EoE (including heartburn, regurgitation, difficulty swallowing, painful swallowing).

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children between the ages of 8-18 years scheduled for endoscopy for clinical indication.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2013-03; Primary Completion 2014-09 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
TEM analysis | at time of sample collection
  Using transmission electron microscopy (TEM), compare mean Dilated Intercellular Space diameter of esophageal epithelium in children with GERD to children with Eosinophilic Esophagitis and normal controls.

SECONDARY OUTCOMES:
pH monitoring | 24 hours
  Evaluate the correlation between mean Dilated Intercellular Spaces diameter and quantitative reflux parameters determined by 24-hour esophageal multichannel intraluminal impedance-pH (MII-pH) monitoring

OTHER OUTCOMES:
Immunoblotting | At time of sample collection
  Evaluate the correlation between mean Dilated Intercellular Spaces diameter and injury to the Intercellular Junctional Complex (IJC) through immunoblotting-based assessment of cleaved versus intact e-cadherin.

CONTACTS AND LOCATIONS:
Overall Officials: Eric H Chiou, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Texas Children's Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Physician Profile — https://www.texaschildrens.org/find-a-doctor/eric-h-chiou-md